CLINICAL TRIAL: NCT06483646
Title: Evaluation of the Stability of Volatile Sulfur Compounds in Gas Samples for Halitosis Diagnosis
Brief Title: Evaluation of the Stability of Sulfur Volatile Compounds From Exhaled Air for Halitosis Diagnosis
Acronym: HALITOSIX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9359
Record Dates: First submitted 2024-06-24; First posted 2024-07-03 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Halitosis
MeSH Terms: conditions — Halitosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Gaseous sampling: — the subject is asked to aspirate the gaseous contents of his oral cavity using a 1ml plastic syringe.

SUMMARY:
Halitosis or bad breath is a problem affecting 30% of the world's population. There are many causes, and oral pathologies, including periodontitis, are the main etiology. In order to make a diagnosis, a clinical interview is necessary to distinguish true halitosis from psychological halitosis. In addition, a measurement of volatile sulfur compounds (VSC), the main molecules involved in bad breath, is necessary. This is done during the consultation by measuring the concentration of VSCs in exhaled air. However, few private practices or hospitals have the necessary equipment to measure VSC. As a result, patients are often obliged to travel long distances to obtain a consultation including this specific VSC analysis. The aim of this study is to evaluate the stability of VSC values obtained in gaseous samples up to 7 days after sampling, in order to assess the clinical relevance of analyzing samples at a distance from sampling. The clinical aim is to determine whether self-sampling by the patient at home and extemporaneous analysis could be considered in the diagnosis of halitosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult, male or female
* Subject affiliated with a social health insurance plan
* Able to understand the objectives and risks of the research and to give dated and signed informed consent
* Subject presenting for consultation for diagnosis and treatment of periodontal pathology

Exclusion Criteria:

* Subject under safeguard of justice
* Subject under guardianship or curatorship
* Pregnancy or breast-feeding
* Impossibility of giving the subject informed information (subject in emergency situation, difficulties in understanding the subject, etc.)
* Subject currently included in another clinical research protocol or in an exclusion period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
H2S measurement | Analysis will be made at Day 0 and Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique dentaire, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No